CLINICAL TRIAL: NCT00630123
Title: Effect of Electroconvulsive Therapy (ECT) and Transcranial Magnetic Stimulation (TMS) on Serum Levels of Brain Derived Neurotrophic Factor in Depressed Patients.
Brief Title: Effect of Electroconvulsive Therapy (ECT) and Transcranial Magnetic Stimulation(TMS) on Brain Derived Neurotrophic Factor (BDNF) in Depressed Patients.
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Roumen Milev, Principal Investigator, Queen's University
Other Study IDs: PSIY-252-06
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum frozen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Electroconvulsive Therapy (ECT): blood sample taken from this group at start and after therapy; subjects not randomized to therapy option.
- 2: Transcranial Magnetic Stimulation (TMS): blood sample taken from this group at start and after therapy; subjects not randomized to therapy option.

SUMMARY:
To investigate the change in brain derived neurotrophic factor (BDNF) between pre and post treatment for patients with depression with either ECT or TMS.

ELIGIBILITY:
Inclusion Criteria:

* MDD or bipolar disorder;
* current depressive episode, ham-d17>17 and ymrs<8;
* recommended to receive ECT or TMS as part of clinical care;
* male/female;
* age 18-65;
* inpatient or outpatient;
* comorbid dysthymic disorder, gad, or social anxiety will be included;
* able to give written consent and agree.

Exclusion Criteria:

* current manic, hypomanic, or mixed episode, ymrs>7;
* current schizophrenia, anorexia, bulimia, substance dependence (current within past 6 months excluding caffeine and nicotine);
* TMS or ECT in the last 3 months;
* any other primary diagnosis;
* uncontrolled medical illness;
* epilepsy or severe personality disorder at the discretion of the investigators;
* 3 weeks prior to first blood test, antidepressants, mood stabilizers, antipsychotics can not be added or increased;
* pregnant women or women of childbearing potential not willing to use appropriate contraception, nursing women;
* known intolerance or lack of response to treatment receiving as judged by the investigator;
* medical conditions that would affect serum levels of BDNF;
* involvement in planning and conduct of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with current major depressive disorder or bipolar depression who are to receive either ECT or TMS.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2006-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Serum levels of BDNF. | pre and post treatment

SECONDARY OUTCOMES:
Correlation between the change in BDNF levels and illness severity after treatment. | pre and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roumen Milev, MD, FRCP(C), Principal Investigator — Queen's University
Locations (1):
- Providence Care Mental Health Services, Kingston, Ontario, Canada